CLINICAL TRIAL: NCT00558766
Title: Motor Cortex Reward Signaling in Parkinson Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080023; 08-N-0023
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-13

CONDITIONS: Parkinson Disease
Keywords: Disruptive Behavior Disorders; Behavior; Gambling; Dopaminergic Mechanisms; Dopamine; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Attention Deficit and Disruptive Behavior Disorders; Behavior; Gambling

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

The brain releases signals to mark rewards for certain behavior. Some medications for Parkinson disease (PD) can cause some patients to engage in compulsive behavior, possibly because the medications affect this reward system.

By using transcranial magnetic stimulation (TMS), researchers can study brain activity when an individual receives a reward.

Objectives:

To learn how the brains of people with PD behave when rewarded.

To learn whether two common Parkinson medications (levodopa and pramipexole) change this behavior.

To compare reward signals in the brains of healthy volunteers with reward signals in the brains of people with PD.

Eligibility:

Women between 50 and 80 years of age and men between 45 and 80 years of age.

Participants will be divided into healthy volunteers and volunteers who have mild to moderate PD.

Design:

Prescreening will consist of a neurological examination and a series of questions about gambling habits and drug and alcohol use.

Participation in a TMS study involving a computer game simulation of a slot machine:

* Before the simulation, participants will receive TMS to establish a baseline response rate.
* During the simulation, participants will play a game in which they will receive real money.

TMS will be administered to each patient under three different conditions:

* TMS administered when patients have not taken any Parkinson medication.
* TMS administered after patients have taken levodopa.
* TMS administered after patients have taken pramipexole....

DETAILED DESCRIPTION:
The role of mesencephalic dopamine neurons in reward processing has been established in primates using electrophysiological techniques and in humans using functional neuroimaging. Their role is thought to be dual: i) they show sustained activity with the expectation of a future reward and ii) a phasic response after reward. Animal data indicate that these neurons, located in the midbrain areas A8-10, behave as a single functional unit when activated. They have rich projections to both the prefrontal and motor cortices where they synapse on interneurons and cortical pyramidal cells, producing primarily inhibition. Though their function is not fully understood, these projections clearly play an important role in motivation and learning. We have recently developed a pair of paradigms to detect a reward related signal in the primary motor cortex, where transcranial magnetic stimulation can be used to measure brief events. So far, we have tested healthy volunteers; we now intend to study Parkinson disease (PD) patients in order to help clarify the role of dopamine in effect of reward. The Parkinson patients will be tested both on and off levodopa/carbidopa and dopamine agonist medications. Our hypothesis is that the dopamine reward related signal will alter level of evocable inhibition in primary motor cortex. Using a behavioral paradigm that deliver intermittent reward, we aim to demonstrate, in treated and untreated PD patients a difference in the amount of cortical inhibition, i) when reward is expected compared to when reward is not expected and ii) after rewarded compared to unrewarded trials. We also aim to demonstrate a difference between their response and that of healthy controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY SUBJECTS:

-Age 45-70 years

PATIENTS:

* Mild-moderate disease (Hoehn and Yahr stage 1-2).
* Age 45-70 yrs

EXCLUSION CRITERIA:

* Pre-menopausal status in women: Preliminary data in healthy, cycling women suggests that the variation in paired-pulse inhibition caused by the menstrual cycle may obscure the change in the response induced by the behavioral task.
* Significant neurological or psychiatric history other than PD
* Exposure to DA agonists within a month of study
* History of habitual gambling, defined as either visiting casinos more than once per month or playing cards for money more than once per week or gambling over the internet more than once per month
* Habitual consumption of more than two drinks a day, marijuana more than once a week or any other illicit drug use within the last three months
* Significant abnormality on neurological examination other than PD related signs
* Metal in the cranial cavity or eye, pacemaker, implanted pumps or stimulators
* Use of non-PD related medications affecting the DA system, such as phenothiazine antihistamines (promethazine), antiemetics or decongestants in the last month

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11-08; Study Completion 2011-06-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Avanzi M, Uber E, Bonfa F. Pathological gambling in two patients on dopamine replacement therapy for Parkinson's disease. Neurol Sci. 2004 Jun;25(2):98-101. doi: 10.1007/s10072-004-0238-z. PMID 15221629
- [Background] Cohen MX, Young J, Baek JM, Kessler C, Ranganath C. Individual differences in extraversion and dopamine genetics predict neural reward responses. Brain Res Cogn Brain Res. 2005 Dec;25(3):851-61. doi: 10.1016/j.cogbrainres.2005.09.018. Epub 2005 Nov 11. PMID 16289773
- [Background] Strobel A, Spinath FM, Angleitner A, Riemann R, Lesch KP. Lack of association between polymorphisms of the dopamine D4 receptor gene and personality. Neuropsychobiology. 2003;47(1):52-6. doi: 10.1159/000068876. PMID 12606846